CLINICAL TRIAL: NCT05843552
Title: Extracellular Vesicles as Potential Biomarkers and Therapeutic Target in Gaucher Disease
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: EV
Record Dates: First submitted 2023-03-31; First posted 2023-05-06 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Gaucher Disease
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — fasting blood samples will be collected. One sample will be collected during first visit for genotyping and will be shipped to commercial lab as per their protocol. Remaining samples will be processed immediately to separate plasma, which will be snap frozen and shipped to University of Minnesota for further analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients with GD
  Interventions: Other: no intervention
- obligate carriers
  Interventions: Other: no intervention
- healthy volunteers
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention, this is an observational study

SUMMARY:
This is an observational study intended to generate preliminary data to understand how lysosomal dysfunction can affect the biogenesis of extracellular vesicles, its content and function. The primary objective of the proposed project is to decipher how extracellular vesicle (EV) biogenesis and its role in intercellular communication can be impaired as a consequence of defects in lysosomal function. Collectively these defects in EV biogenesis and function can contribute to the neuroinflammation observed in lysosomal storage diseases. Since EVs can cross the blood-brain barrier, their characterization may be valuable in identifying novel biomarkers. In the presence of a GBA1 mutation, the decrease in GCase activity will lower overall lysosome function and increase the secretion of EVs. Further, there will be differences in EV size, its cargo including lipids, RNA and proteins and their aggregates. In comparison to healthy controls, EVs isolated from patients with Gaucher disease (GD) and GBA1 carriers is hypothesized to show significant differences in terms of its characteristics and content, which can contribute to our understanding of the link between lysosomes and neurological disease.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-80yrs
* Restricted to participants who are untreated, obligate carriers and healthy controls.
* Participants with GD should have confirmed GD diagnosis, mutation confirmed for carriers and healthy controls confirmed to have no GBA1 mutation by gene sequencing.

Exclusion Criteria:

* Exclude participants who have any hematological malignancy or other uncontrolled comorbid conditions.
* Exclude participants who are currently on therapy for their GD
* Exclude participants who have any hematological malignancy or other uncontrolled comorbid conditions.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with GD (n=10 untreated), obligate carriers (n=10) and healthy volunteers (frequency matched for age and gender; n=10) for this study. In the next phase of this project, we will examine the effect of GD treatment on EV characteristics by focusing on patients who are currently being treated and compare various therapies and correlate it with established biomarkers.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-04-30 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
EVs quantity | baseline
  Examine EV quantities isolated from plasma samples collected from patients with GD and carriers and compare to healthy individuals.
EVs quantity | 3months
  Examine EV quantities isolated from plasma samples collected from patients with GD and carriers and compare to healthy individuals.
EVs size | baseline
  Examine EV sizes isolated from plasma samples collected from patients with GD and carriers and compare to healthy individuals.
EVs size | 3months
  Examine EV sizes isolated from plasma samples collected from patients with GD and carriers and compare to healthy individuals.
EVs content | baseline
  Examine contents in vesicles isolated from plasma samples collected from patients with GD and carriers and compare to healthy individuals.
EVs content | 3months
  Examine contents in vesicles isolated from plasma samples collected from patients with GD and carriers and compare to healthy individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Reena Kartha, PhD, MS, Principal Investigator — University of Minnesota; Subbaya Subramanian, PhD, MS, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States